CLINICAL TRIAL: NCT05609045
Title: A Phase 1, Randomised, Double-blinded, Placebo-controlled, Dose-escalation Study to Evaluate the Safety and Immunogenicity of RH109 as Booster for Healthy Adults Who Have Received Homologous or Heterologous Vaccination With 3 Doses of COVID-19 Inactivated and/or mRNA Vaccine(s)
Brief Title: A Phase 1, Randomised, Double-blinded, Placebo-controlled, Dose-escalation Study to Evaluate the Safety and Immunogenicity of RH109 as Booster
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: business strategy adjustment
Sponsor: Wuhan Rhegen Biotechnology Co., Ltd. (Industry)
Collaborators: Shenzhen Rhegen Biotechnology Co.,Ltd. (Industry); Wuhan Recogen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RH109 CT HK01
Record Dates: First submitted 2022-10-28; First posted 2022-11-08 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test product group (Experimental)
  Interventions: Biological: Lyophilized COVID-19 mRNA Vaccine
- placebo group (Placebo Comparator)
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Biological: Lyophilized COVID-19 mRNA Vaccine — RH109 is a mRNA-based vaccine encoding the N-Terminal Domain (NTD) - Receptor Binding Domain (RBD) derived from Spike (S) protein of SARS-CoV-2 Omicron variant.
  Arms: test product group
Drug: Sodium chloride — 0.9% sodium chloride
  Arms: placebo group

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, dose-escalation study to valuate the safety and immunogenicity of RH109 as booster at 2 dose levels for ealthy adults who have received homologous or heterologous vaccination with 3 doses of COVID-19 inactivated and/or mRNA vaccine(s).

The purpose of this study is to evaluate the safety and immunogenicity of RH109 as booster for healthy adults who have received homologous or heterologous vaccination with 3 doses of COVID-19 inactivated and/or mRNA vaccine(s).

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible for inclusion in this study if all of the following criteria are met:

1. Informed Consent: The subject (or the subject's legally acceptable representative, if applicable) must be capable of giving written informed consent and, prior to the commencement of any study-specific procedure, must sign an ICF indicating the consent on the subject's voluntary participation in the study and compliance with the requirements and restrictions listed on the ICF.
2. Vaccination Status: The subject must have received homologous or heterologous vaccination with 3 doses of COVID-19 inactivated and/or mRNA vaccine(s) recognized by the local health authorities, with the last dose completed at least 90 days prior to IMP vaccination.
3. Gender and Age: Male or female, at the age of ≥ 18 and ≤ 80 on the day of signing the ICF.
4. Body Weight and BMI: Body weight ≥ 45 kg and BMI ≥ 18.5 kg/m2 and < 30 kg/m2 at screening and baseline.
5. Medical Conditions or Diagnoses: Existence of all of the following medical conditions or diagnoses:

   1. Generally in good health with no clinically significant abnormality, as determined by medical history, physical examination, 12-lead ECG and clinical laboratory tests at screening and baseline;
   2. Normal vital signs at screening and baseline, as defined by:

      * Body (tympanic) temperature ≤ 37.5°C;
      * Resting pulse rate ≥ 50 and ≤ 100 bpm; and
      * DBP ≥ 50 and ≤ 90 mmHg and SBP ≥ 90 and ≤ 140 mmHg.
6. Avoidance of Pregnancy: Willingness and agreement to undertake measures to confirm the subject's non-childbearing potential or avoid pregnancy of the subject or the subject's sexual partner(s) as detailed below:

   1. A female subject who declares menopause must (i) confirm that she has not experienced a menstrual period for at least 12 consecutive months; and (ii) be willing to receive a FSH test to confirm her postmenopausal status;
   2. A female subject who declares completion of surgical sterilization (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal occlusion or ligation) must be able to provide valid medical evidence or permit access to the relevant medical records;
   3. A female subject who is a woman of childbearing potential (WOCBP) must be willing and agree to remain abstinent or practise at least one effective contraceptive method from at least 30 days prior to the day of IMP vaccination and for 60 days after IMP vaccination;
   4. A male subject (i) who is sexually active with a WOCBP (except who is permanently sterile by bilateral orchiectomy or vasectomy) must be willing and agree to remain abstinent or practise at least one effective contraceptive method from the day of IMP vaccination and until 60 days after IMP vaccination; and (ii) must be willing and agree to refrain from sperm donation during the aforesaid period.
7. Breastfeeding: A female subject must be willing and agree to avoid engagement in breastfeeding at any time from the day of IMP vaccination until 60 days after IMP vaccination.
8. Blood Donation: Willingness and agreement to avoid blood donation from screening to the end of the period of participation in this study.

Exclusion Criteria:

A subject is excluded from this study if any of the following criteria applies:

1. Medical History: History of any of the following diseases or conditions:

   1. COVID-19;
   2. SARS;
   3. Any significant respiratory diseases (e.g. COPD, asthma);
   4. Any significant cardiovascular disease (e.g. angina, cardiac arrhythmias);
   5. Blood dyscrasias or any significant disorder of coagulation;
   6. Any chronic liver disease (e.g. autoimmune hepatitis and cirrhosis);
   7. Any chronic infection (e.g. hepatitis B, hepatitis C and HIV);
   8. Any malignant neoplastic disease;
   9. Encephalopathy, neuropathy or unstable central nervous system (CNS) pathology;
   10. Any psychiatric disorder, psychotic disorder, major affective disorder or suicidal ideation;
   11. Any immunodeficiency or autoimmune disease;
   12. Any severe allergic reaction (e.g. anaphylaxis) to any vaccine or substance, which requires hospitalization or emergency medical care;
   13. History of alcohol or illicit drug abuse, or used any illicit drug within 6 months prior to screening.
2. Medical Conditions or Diagnoses: Existence of any of the following medical conditions or diagnoses:

   1. Positive serum pregnancy test at screening or positive urine pregnancy test at baseline (only for WOCBP);
   2. Serum FSH test result at screening indicating a postmenopausal status (only for women declaring menopause for at least 12 consecutive months prior to screening);
   3. IgE level > 1,000 IU/ml at screening;
   4. Positive Anti-N IgG test result at screening;
   5. Positive SARS-CoV-2 test result in deep throat saliva (DTS) within 4 days prior to the day of vaccination;
   6. Positive HIV test result at screening;
   7. Positive HBsAg test result at screening;
   8. Positive HCV antibody test result at screening;
   9. Positive urine drug screen test result or positive blood alcohol test result at screening or baseline;
   10. Clinically significant abnormality of T3, T4 or TSH at screening;
   11. Clinically significant abnormality of PT (INR) or aPTT at screening.
3. Prior/Concomitant Interventions: Use of or undergoing any of the following prior or concomitant medications, therapies or interventions:

   1. Any COVID-19 or coronavirus vaccine at any time prior to IMP vaccination (except the inactivated and mRNA vaccines recognized by the local authorities of the respective study sites), or planned use of any such vaccine throughout the study;
   2. Any vaccine other than COVID-19 or coronavirus vaccines within 28 days prior to IMP vaccination, or planned use of any such vaccine up to 28 days after IMP vaccination;
   3. Any immune-modifying medication/therapy (e.g. immunomodulator and immunosuppressant) within 6 months prior to IMP vaccination, or planned use of any such medication/therapy throughout the study;
   4. Any blood product (including blood transfusion) or immunoglobulin within 4 months prior to IMP vaccination, or planned use of any such therapy throughout the study;
   5. Any anticoagulation medication within 28 days prior to IMP vaccination, or planned use of any such medication up to 28 days after IMP vaccination;
   6. Any psychotropic medication within 28 days prior to IMP vaccination, or planned use of any such medication up to 28 days after IMP vaccination;
   7. Any prescription or over-the-counter medication within 7 days prior to IMP vaccination, unless with the investigator's approval;
   8. Donated ≥ 450 mL of blood within 28 days prior to IMP vaccination.
4. Prior/Concurrent Clinical Study: Prior or concurrent participation in any other clinical study, including:

   1. Prior or current participation in another COVID-19 vaccine study;
   2. Prior participation in any interventional clinical study and use of any investigational intervention within 30 days prior to IMP vaccination;
   3. Concurrent participation or plan for participation in another interventional clinical study during participation in this study.
5. Other Significant Medical Conditions: Any clinically significant concomitant disease or condition that, in the reasonable opinion of the investigator, may interfere with the subject's participation in this study or pose an unacceptable safety risk for the subject's participation in this study.
6. Special Condition: Existence of the following special condition:

   1. Planned to travel overseas at any time during the period from screening to Day 90(±7) visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reactogenicity | Day0 to Day7
  Incidence of any solicited local events (pain, tenderness, redness, warmth, itch, welling, induration) and solicited systemic events (fever, headache, malaise, fatigue, yalgia, joint pain, nausea, vomiting, diarrhea, loss of appetite, chills) after IMP vaccination.
Unsolicited Treatment Emergent Adverse Events (TEAEs): | Day0 to Day28
  Incidence of unsolicited TEAEs after IMP vaccination.
Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs): | Day0-Day90
  Incidence of AESIs and SAEs after IMP vaccination.

SECONDARY OUTCOMES:
geometric mean titre (GMT) | Day 7, Day 21, Day 28, Day 60 and Day 90
  GMT of neutralizing antibodies against Omicron, Wild-type or other selected variants
geometric mean increase (GMI) | Day 7, Day 21, Day 28, Day 60 and Day 90
  GMI of anti-Omicron neutralizing antibody, anti-Omicron IgG antibodies
geometric mean concentration (GMC) | Day 7, Day 21, Day 28, Day 60 and Day 90
  GMC of anti-Omicron IgG antibodies
seroconversion rate (SCR) | Day 7, Day 21, Day 28, Day 60 and Day 90
  SCR of anti-Omicron neutralizing antibody, anti-Omicron IgG antibody
T-Cell Responses | Day 7, Day 21, Day 28, Day 60 and Day 90
  Median T-cell responses

IPD SHARING:
Plan to Share IPD: No